CLINICAL TRIAL: NCT01124942
Title: MGuard vs bAre-metal Stents Plus Manual Thrombectomy in Real World STEMI Patients: a Prospective Multicenter Randomized Trial
Brief Title: MGuard Stent in ST-elevation Myocardial Infarction
Acronym: GUARDIAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giovanni Esposito, Cardiologist, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA116/09
Record Dates: First submitted 2010-04-08; First posted 2010-05-18 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: ST-elevation Myocardial Infarction; Thrombus; Stents
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MGuard (Experimental): MGuard net protective stent, investigational device
  Interventions: Device: MGuard net protective coronary stent
- BMS plus thrombectomy (Active Comparator): Bare-metal stent plus manual thrombectomy device
  Interventions: Device: Bare-metal stent and manual thrombectomy device

INTERVENTIONS:
Device: MGuard net protective coronary stent — It is a new closed-cell design stent concept. with an ultra-thin flexible polyethylene terephthalate (or Dacron) mesh sleeve, anchored to the external surface of the struts. This net (string diameter 10-22 μm) minimally affects stents' trackability and deliverability. During stent deployment, the net stretches and slides over the expanding stent struts, trapping the thromboembolic debris underneath the fiber net.
  Other Names: MGuard net protective stent
  Arms: MGuard
Device: Bare-metal stent and manual thrombectomy device — Manual thrombectomy device as an adjunctive strategy for conventional stenting with a bare-metal stent
  Arms: BMS plus thrombectomy

SUMMARY:
The Investigators will test the hypothesis that MGuard net protective stent, the investigational device, would be superior to conventional revascularization strategy (i.e. bare-metal stenting plus manual thrombectomy), for STEMI patients undergoing urgent percutaneous coronary interventions.

DETAILED DESCRIPTION:
Embolization of thrombotic debris still represents a complication for ST-elevation myocardial infarction (STEMI) patients undergoing percutaneous coronary interventions (PCI).

Distal embolization may decrease coronary and myocardial reperfusion after PCI in STEMI setting.

Unfortunately, intracoronary filters present several important limitations limiting their use and their efficacy especially in presence of huge amount of thrombus. In this respect, recent trials investigated whether a default manual thrombectomy strategy before stenting would ameliorate angiographic as well as clinical outcomes for STEMI patients undergoing percutaneous revascularization.

Of note, the most of embolization occurs when guidewire, and thrombectomy device cross the thrombus, and after the stent has been implanted as a consequence of plaque prolapse through the stent struts.

MGuard net protective stent, the investigational device, is a bare-metal stent covered with a ultra-thin flexible polyethylene terephthalate (or Dacron) mesh sleeve, that is anchored to the external surface of the struts. This biocompatible fiber net (string diameter 10-22 μm) has minimal effects on the stents' trackability and deliverability. During stent deployment, the net stretches and slides over the expanding stent struts, trapping the thromboembolic debris underneath the fiber net and isolating the prothrombotic intima components from the blood stream.

This protocol will test the hypothesis that MGuard stent would be superior to conventional revascularization strategy (i.e. bare-metal stenting plus manual thrombectomy), for STEMI patients undergoing urgent PCI in terms of angiographic as well as clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18-year-old patients, willing to participate the study, after informed consent signature
* Female not pregnant or potentially child-bearing
* > 1 mV ST segment elevation in two or more contiguous leads
* Acute MI lasting more than 30 minutes and less than 12 hours
* De novo acute MI
* Infarct related artery reference vessel diameter >/= 2.5 mm
* Patient suitable for stenting according to vessel and lesion features

Exclusion Criteria:

* Dual antiplatelet therapy contraindication
* Ischemic stroke less than 30 days or previous haemorrhagic stroke
* WBC count less than 1000 per mm3;
* Platelet count less than 50.000 per mm3
* Life expectancy less than 1 year
* Cardiogenic shock at admission
* Previous stented infarct related artery
* Stent thrombosis as the responsible for current STEMI
* Inability to identify infarct related artery
* True bifurcation lesion, or lesion near a side branch with a reference vessel diameter >/= 2.5 mm that could be diseased after stenting procedure
* LBBB
* Definitive pacing (or ECG abnormalities precluding ST-segment resolution evaluation
* Participation other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2013-03-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with Myocardial Perfusional Blush Grade 2-3 | 30 minutes after revascularization
  Myocardial Perfusional Blush Grade 2-3 at the end of the procedure

SECONDARY OUTCOMES:
Number of MACE | 1 month
  Number of Major Adverse Cardiovascular Events experienced among study population, including: cardiac death, myocardial infarction, target vessel failure.
Complete ST-segment resolution | 60 minutes after revascularization
  Complete (>70%) ST-segment resolution at 60 minutes post-revascularization
Thrombolysis in myocardial infarction antegrade coronary flow | 30 minutes after revascularization
  TIMI coronary flow at the end of the procedure
Corrected TIMI Frame count | 30 minutes after revascularization
  Corrected TIMI Frame count at the end of the procedure
Infarct related area reduction and left ventricular ejection fraction recovery | 6 months
  Six-month infarct related area reduction and left ventricular ejection fraction recovery as compared with infarct related area and and left ventricular ejection fraction at admission.
Procedural device performance | 60 minutes after revascularizationl
  Device performance evaluated during the procedure in terms of pushability, trackability, crossability and deliverability
Number of MACE | 6 months
  Number of Major Adverse Cardiovascular Events experienced among study population, including: cardiac death, myocardial infarction, target vessel failure.
Number of MACE | 12 months
  Number of Major Adverse Cardiovascular Events experienced among study population, including: cardiac death, myocardial infarction, target vessel failure.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Piscione, Associate Professor, Study Chair — Federico II University of Naples
Locations (1):
- Federico II University of Naples, Naples, Italy

REFERENCES:
- [Background] Piscione F, Danzi GB, Cassese S, Esposito G, Cirillo P, Galasso G, Rapacciuolo A, Leosco D, Briguori C, Varbella F, Tuccillo B, Chiariello M. Multicentre experience with MGuard net protective stent in ST-elevation myocardial infarction: safety, feasibility, and impact on myocardial reperfusion. Catheter Cardiovasc Interv. 2010 Apr 1;75(5):715-21. doi: 10.1002/ccd.22292. PMID 19937780
- [Background] Rapacciuolo A, D'andrea C, Maresca G, di Pietro E, Piscione F, Chiariello M. Multiple MGuard stent implantation to treat massive right coronary artery dissection during primary coronary angioplasty. J Cardiovasc Med (Hagerstown). 2011 May;12(5):356-60. doi: 10.2459/JCM.0b013e328334092d. PMID 20093945